CLINICAL TRIAL: NCT05195931
Title: Factors Affecting Resting and Exertional Cardiac Output and HVAD Flow Among Patients With Advanced Heart Failure - A PILOT STUDY
Brief Title: Cardiac Output in Heart Failure Patients With Mechanical Pumps
Status: Terminated | Type: Observational
Why Stopped: Withdrawal of funding by study sponsor
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2143
Record Dates: First submitted 2021-06-18; First posted 2022-01-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure, Systolic; Mechanical Circulatory Support; Cardiovascular Hemodynamics
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preload and Afterload: 10 participants with heart failure who are supported by LVADs will undergo hemodynamic monitoring and observation while undergoing changes in preload (head-up tilt and saline infusion), and afterload (nitroprusside and phenylephrine infusion).
  Interventions: Diagnostic Test: preload challenge; Diagnostic Test: afterload challenge
- Contractility: 10 participants with heart failure who are supported by LVADs will undergo hemodynamic monitoring and observation while undergoing changes in contractility with adjustments in heart rate (by adjusting pacemaker), dobutamine infusion, and during exercise.
  Interventions: Diagnostic Test: contractility assessment

INTERVENTIONS:
Diagnostic Test: preload challenge — reduction in preload by head-up tilt and increase in preload with saline infusion
  Groups: Preload and Afterload
Diagnostic Test: afterload challenge — reduction in afterload with nitroprusside and increase in afterload with phenylephrine
  Groups: Preload and Afterload
Diagnostic Test: contractility assessment — heart rate changes will be made by increasing heart rate with external pacemaker/defibrillator. Contractility will be adjusted by dobutamine infusion. Patients will exercise at a constant pump speed and also with pump speed increases.
  Groups: Contractility

SUMMARY:
This study will be looking at how cardiovascular hemodynamics, including cardiac output and flow through a left ventricular assist device (LVADs), change in response to alterations in preload, afterload, and contractility, and also during exercise, in humans with heart failure who are supported by LVADs.

DETAILED DESCRIPTION:
Heart failure is a devastating disease, which affects approximately 6 million individuals in the USA alone. Five-year survival among all-comers with HFrEF is ~50%, and there are associated reductions in functional capacity and health-related quality-of-life (HRqOL). While guideline-directed medical therapy such as beta-blockers, angiotensinogen converting enzyme inhibitors, mineralocorticoid receptor antagonists and angiotensin receptor-neprilysin inhibitors improve survival, HRqOL and functional capacity, many patients progress to end-stage, advanced HFrEF, which has a five-year survival of only to 20% and is associated with reductions in functional capacity and HRqOL. While orthotopic heart transplantation is the gold-standard treatment for advanced HFrEF, only approximately 3,000 donor organs are available per year in the USA, and approximately 5,000 per year worldwide. As such, demand outweighs supply since estimates are that at least 50,000 individuals worldwide are candidates for transplant or suffer from severe HFrEF and are transplant ineligible for a variety of reasons (e.g. uncontrolled diabetes mellitus or peripheral vascular disease, or diagnosis of cancer within the past 5 years). To remedy this disparity, LVADs have emerged as an attractive alternative and are used as either a bridge-to-transplantation to stabilize and support patients until transplantation is possible, or as destination-therapy for transplant-ineligible patients. HFrEF patients frequently suffer from elevated cardiac filling pressures and reduced cardiac output (Qc) under resting conditions. LVADs normalize these hemodynamic abnormalities - at least under resting conditions - through a rotating impeller that propels blood from the left ventricle (LV) into the ascending aorta (figure 1). Total Qc is therefore determined by: 1) the LVAD, which provides the bulk of flow to the body during resting conditions; and 2) the native heart, which can still provide blood to the body by expulsion of blood through the aortic valve as the heart contracts.

Heart failure patients suffer from persistent heart failure symptoms, and impairments in functional capacity, following LVAD implantation. It has previously been demonstrated that LVAD patients have severely reduced functional capacity, as measured by serial assessments of maximal oxygen uptake (VO2Max), greater than one year following device implantation.27 Specifically, VO2Max, when assessed before LVAD implantation, 3-6 months, 1 year, and greater than 1 year following device implantation, remains below 14ml/kg/min. Submaximal exercise, measured by six-minute hall walk (6MHW) scores, improves modestly following device implantation, but on average, remains severely reduced at approximately 300-350m, and similar to VO2Max values observed in these patients, falls within a range that is observed among patients with advanced HFrEF. About half of patients report persistence of HFrEF-related symptoms 6-12 months following device implantation. These persistent reductions in VO2Max, 6MHW, and HRqOL assessments all indicate that LVAD patients suffer from persistent heart failure, which manifests with attempts to exercise. For example, HFrEF patients are considered to be eligible for a heart transplantation when their VO2Max falls below 12-14ml/kg/min.

Impairments in HRqOL and functional capacity result from an inability of the LVAD to improve cardiovascular hemodynamics during exercise. To understand how LVADs influence cardiac filling pressures at rest and during exercise, we previously evaluated patients prior to, and following LVAD implantation by invasive cardiopulmonary exercise testing (CPET) with Swan-Ganz catheterization during upright cycle ergometry prior to and following LVAD implantation (COMIRB #16-1635). In this study (figure 2), three visits were completed: 1) Visit 1: baseline exercise assessment four weeks before LVAD implantation. 2) Visit 2: post-LVAD exercise assessment with patient exercising at constant LVAD pump speed. 3) Visit 3: post-LVAD exercise assessment but with stepwise increases in LVAD rotor speed during exercise, to determine whether additional flow through device improves exercise capacity. Several novel insights resulted from this work (figure 2):

1. Cardiopulmonary performance remains severely limited following device implantation. Compared to pre-LVAD CPET (visit 1), there is no improvement in VO2Max following LVAD implantation when patients exercise to volitional exhaustion at either a constant pump speed (visit 2), or with stepwise increases in pump speed (visit 3).
2. LVAD flow increases minimally during exercise. Regardless of whether LVAD patients exercise at a constant pump speed or with stepwise increases in speed, LVADs can only increase flow by approximately 1L/min above resting levels. As such, cardiac output during exercise - and hence, VO2Max - is determined by contractile reserve of the native ventricle, as opposed to the LVAD itself.
3. Exertional pulmonary arterial and cardiac filling pressures do not improve following LVAD implantation. Pre-implantation exertional filling pressures (visit 1) are severely elevated in the setting of advanced HFrEF, and interestingly, there is no substantive improvement following device implantation when exercising at a fixed LVAD speed or with stepwise increases in pump speed.

There is a paucity of data regarding the impact of changes in hemodynamics on LVAD function in the human body. The effects of alterations in afterload, preload and contractility in the normal heart are well described. For example, left ventricular (LV) pressure-volume analysis (the gold-standard metric of describing ventricular function) indicates that there is an inverse relationship between afterload and Qc, such that increases in afterload lead to reductions in Qc, and vice versa. However, preload is directly related to Qc, such that increases in cardiac preload lead to a rise in Qc through the Frank-Starling mechanism. In vitro studies of LVADs suggest that - at least in the controlled environment of a "mock-loop" (figure 3), LVADs have a reduced preload sensitivity than the normal heart. For example, LVAD preload sensitivity is approximately half the levels observed in the normal heart (LVAD v. heart, 0.105±0.092 v. 0.213±0.003 L/min/mmHg). However, similar mock-loop studies suggest that LVADs have a much higher afterload sensitivity - approximately three times - that of the normal heart (LVAD v. heart 0.09±0.034 v. 0.03±0.01 L/min/mmHg). The main limitation with these mock-loop studies, however, is that for variables such as preload and afterload, which all contribute to changes in flow - these variables are changed in isolation (e.g. increasing preload while holding afterload constant), whereas in the human body, all variables change simultaneously during activity. As such, these mock-loop studies do not adequately describe - or explain, LVAD flow behavior during exercise, where preload increases, afterload decreases, and contractility increases, but LVAD flow increases minimally or not at all (point #2 above). It has previously been emphasized that a detailed understanding of exercise physiology in this patient population is necessary to improve HRqOL and exercise tolerance in this patient population. Therefore, the primary objective of this study is to evaluate LVAD performance in response to alterations in loading conditions (preload, afterload, contractility) in HFrEF patients supported by these devices, and characterize the determinants of LVAD flow and Qc during activity/exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years of age or greater;
2. Clinically stable, ambulatory outpatients with HVAD who are fully recovered from surgical implantation.

Exclusion Criteria:

1. Confirmed or suspected device malfunction (e.g. pump thrombus, LVAD-related infection);
2. Clinical instability, defined as hypotension (mean arterial pressure < 60mmHg and symptomatic, as measured in the advanced heart failure LVAD clinic), or hypertension (mean arterial pressure > 90mmHg); patients with refractory heart failure symptoms with New York Heart Association functional classification IIIB or IV symptoms;
3. any chronic illness which would render the patient unable to complete the protocol as described, including but not limited to: moderate-severe osteoarthritis, severe pulmonary disease requiring supplemental oxygen, uncontrolled hypertension, a high baseline HVAD pump speed above 2860RPM (exercise protocol requires increasing pump speed by up to 240 RPM);
4. chronic kidney disease with a glomerular filtration rate < 30ml/min/1.73m2;
5. absence of a pacemaker-defibrillator (necessary for pacing assessment as described below);
6. individuals with clinical evidence of right ventricular (RV) dysfunction/failure, defined as moderate-severe hypervolemia on physical examination with elevated jugular venous pressure greater than 10cmH20, imaging evidence of severe RV dysfunction by imaging assessment or tricuspid annular plane systolic excursion < 17mmHg, or use of outpatient inotropes for known history of RV dysfunction.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced heart failure who are supported by an LVAD
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
cardiac output | 5 minutes
  cardiac output from Swan-Ganz catheter

SECONDARY OUTCOMES:
mean arterial pressure | 5 minutes
  mean arterial pressure during hemodynamic testing
LVAD flow | 5 minutes
  LVAD flow from device programmer during hemodynamic testing
right atrial pressure | 5 minutes
  right atrial pressure during hemodynamic testing
mean pulmonary arterial pressure | 5 minutes
  mean pulmonary arterial pressure during hemodynamic testing
pulmonary capillary wedge pressure | 5 minutes
  pulmonary capillary wedge pressure during hemodynamic testing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Snschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No